CLINICAL TRIAL: NCT00587431
Title: Docetaxel With Rapid Hormonal Cycling as a Treatment for Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-076; NCT00070369 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Docetaxel; 03-076
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Gonadotropin-Releasing Hormone; Leuprolide; Injections, Intramuscular; Testosterone; Docetaxel

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: GnRh (Leuprolide); Drug: Testosterone Gel; Drug: Docetaxel
- 2 (Active Comparator)
  Interventions: Drug: GnRh (Leuprolide); Drug: Testosterone Gel

INTERVENTIONS:
Drug: GnRh (Leuprolide) — Leuprolide LUPRON
  Other Names: 22.5 mg intramuscular injection
Drug: Testosterone Gel — Starting during week 3 (day 19) of cycle 1, 7.5G applied topically daily for 3 days (applied at approximately 9p)
  Other Names: AndroGel
Drug: Docetaxel — 70 mg/m2 given on day o1 of each 3 week cycle
  Other Names: Taxotere
  Arms: 1

SUMMARY:
We postulate that multiple apoptototic events are indusce through testosterone depletion and repletion with taxotere given in conjunction with androgen withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate adenocarcinoma histologically confirmed at MSKCC or SKCCC.
* Patient must have a serum testosterone > 180 ng/dl.
* Karnofsky performance status (KPS)>_70%.
* Patients must have adequate organ function as defined by the following
* laboratory criteria:
* WBC >_ 3500/mm3
* ANC >_1500/mm3
* Platelet count >100,000/mm3
* Hemoglobin >8.0g/dL
* Creatinine <1.6mg/dl
* Total Bilirubin WNL (unless due to Gilbert's disease and other LFTs are WNL)
* SGOT and SGPT If alkaline phosphatase is _< 2.5 x ULN, any elevations in
* AST/ALT; OR if AST/ALT is _<1.5 x ULN, any elevation in alkaline phos
* Prior hormonal therapy is allowed as:

  1. Neoadjuvant treatment prior to radiation therapy or radical pmstatectomy, provided that the total duration of therapy does not exceed 6 months (Proscar is not considered a hormone therapy).
  2. One cycle of intermittent therapy up to a maximum exposure of 6 months (Proscar is not considered a hormone therapy).
* Patients must be at least 18 years of age.
* Patients must have signed an informed consent document stating that they understand the investigational nature of the proposed treatment

Exclusion Criteria:

* Clinically significant cardiac disease (New York Heart Association Class III/IV), or severe debilitating pulmonary disease.
* Uncontrolled serious active infection.
* Anticipated survival of less than 3 months.
* Active CNS or epiduraltumor
* Inability or unwillingness to comply with the treatment protocol, follow-up, or research tests
* Peripheral neuropathy >_ grade 3.
* Patients with a history of severe hypersensitivity reaction to drugs formulated with polysorbate 80.
* Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 6 months after completion of the treatment.
* Prior chemotherapy
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, St. Johns's Wort (hypericum perforatum) and ketoconazole is prohibited.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Rathkopf, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: 07/08/2003
  Protocol Closed to Accrual: 02/28/2006
  Primary Completion Date: 02/26/2008
  Recruitment Location is the Medical Clinic
Groups:
- Lupron and Docetaxel (75mg/m2) and Testosterone for 7 Days: GnRh (Leuprolide): Leuprolide LUPRON
  Docetaxel: 75 mg/m2 given on day 1 of each 3 week cycle
  Testosterone Gel: Starting during week 3 (day 19) of cycle 1, 7.5G applied topically daily for 7 days
- Lupron and Docetaxel (70 mg/m2) and Testosterone for 3 Days: GnRh (Leuprolide): Leuprolide LUPRON
  Docetaxel: 70 mg/m2 given on day 1 of each 3 week cycle
  Testosterone Gel: Starting during week 3 (day 19) of cycle 1, 7.5G applied topically daily for 3 days
Period: Overall Study
Arm/Group | Lupron and Docetaxel (75mg/m2) and Testosterone for 7 Days | Lupron and Docetaxel (70 mg/m2) and Testosterone for 3 Days
Started | 63 | 39
Completed | 62 | 38
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lupron and Docetaxel (75mg/m2) and Testosterone for 7 Days | Lupron and Docetaxel (70 mg/m2) and Testosterone for 3 Days | Total
Number analyzed (Participants) | 63 | 39 | 102
Age, Continuous [Median (Standard Deviation); unit: years] | 65 (25.45584412) | 58.5 (26.1629509) | 61.5 (30.40559159)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 26 | 69
  >=65 years | 20 | 13 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 63 | 39 | 102
Region of Enrollment [Number; unit: participants]
  United States | 63 | 39 | 102

OUTCOME MEASURES:

1. Primary Outcome: PSA of <_ 0.05 ng/ml After Radical Prostatectomy or Radiation Therapy and PSA <_ 2.0 ng/ml for Patients With Clinical Metastases Without Prior Definitive Therapy
Time Frame: Conclusion of the study (at 6 months then at 18 months post-treatment)
Measure: Number; unit: participants
Groups:
- Lupron + Docetaxel (75mg/m2) +Testosterone (RISING PSA); Lupron + Docetaxel (75mg/m2) + Testosterone for (Metastatic): GnRh (Leuprolide): Leuprolide LUPRON
  Docetaxel: 75 mg/m2 given on day 1 of each 3 week cycle
  Testosterone Gel: Starting during week 3 (day 19) of cycle 1, 7.5G applied topically daily for 7 days
- Lupron +Docetaxel (70 mg/m2) +Testosterone (RISING PSA): GnRh (Leuprolide): Leuprolide LUPRON
  Docetaxel: 70 mg/m2 given on day 1 of each 3 week cycle
  Testosterone Gel: Starting during week 3 (day 19) of cycle 1, 7.5G applied topically daily for 3 days
- Lupron + Docetaxel (70 mg/m2) + Testosterone (Metastatic): (Metastatic) GnRh (Leuprolide): Leuprolide LUPRON
  Docetaxel: 70 mg/m2 given on day 1 of each 3 week cycle
  Testosterone Gel: Starting during week 3 (day 19) of cycle 1, 7.5G applied topically daily for 3 days
Arm/Group | Lupron + Docetaxel (75mg/m2) +Testosterone (RISING PSA) | Lupron + Docetaxel (75mg/m2) + Testosterone for (Metastatic) | Lupron +Docetaxel (70 mg/m2) +Testosterone (RISING PSA) | Lupron + Docetaxel (70 mg/m2) + Testosterone (Metastatic)
Number analyzed (Participants) | 25 | 37 | 17 | 21
participants
  at 6 months post-treatment | 9 | 14 | 13 | 12
  at 18 months post-treatment | 0 | 0 | 3 | 2

2. Secondary Outcome: The Effects of Testosterone Administration on Docetaxel Pharmacokinetics.
Description: Docetaxel Pharmacokinetic parameters for cycles 1 and 2.
Time Frame: at Cycle 1 and 2
Population: A population pharmacokinetic model was fit to the data from all individuals simultaneously using a non-linear mixed effects modeling. This was performed using NONMEM. The NONMEM model accounts for between-patient, between-course, and residual variability (random effects) as well as parameter differences predicted by covariates (fixed effects).
Measure: Mean (Standard Deviation); unit: L/hr
Groups:
- All Participants: All participants
Arm/Group | All Participants
Number analyzed (Participants) | 102
L/hr
  Docetaxel clearance (Cycle 1) | 23.9 (12.1)
  Docetaxel clearance (Cycle 2) | 23.6 (7.43)

ADVERSE EVENTS:
Time Frame: From the start of treatment through 30 days after completing treatment
Arm/Group | Lupron and Docetaxel (75mg/m2) and Testosterone for 7 Days | Lupron and Docetaxel (70 mg/m2) and Testosterone for 3 Days
Serious Adverse Events (participants affected / at risk) | 36/63 | 8/39
Other Adverse Events (participants affected / at risk) | 63/63 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lupron and Docetaxel (75mg/m2) and Testosterone for 7 Days (N=63) | Lupron and Docetaxel (70 mg/m2) and Testosterone for 3 Days (N=39)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 4 (4)
Fever (General disorders) | 2 (2) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (18) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophil count decrease (Investigations) | 27 (49) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hyperhidrosis (excessive perspiration) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lupron and Docetaxel (75mg/m2) and Testosterone for 7 Days (N=63) | Lupron and Docetaxel (70 mg/m2) and Testosterone for 3 Days (N=39)
Fatigue (General disorders) | 57 (57) | 38 (38)
Hot flashes (Vascular disorders) | 41 (41) | 30 (30)
Neuropathy (Nervous system disorders) | 26 (26) | 25 (25)
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 (9) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 41 (41) | 27 (27)
Hyperglycemia (Metabolism and nutrition disorders) | 54 (54) | 38 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes